CLINICAL TRIAL: NCT06537284
Title: Randomized Controlled Trial of Imagery Rescripting With and Without Reconsolidation Disruption
Brief Title: Comparison of Imagery Rescripting With and Without Reconsolidation Disruption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaroslaw Michalowski (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Sponsor-Investigator, Jaroslaw Michalowski, Professor, University of Social Sciences and Humanities, Warsaw
Organization: University of Social Sciences and Humanities, Warsaw (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: SONATA_BIS_JM2019
Record Dates: First submitted 2024-07-22; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Fear of Failure
Keywords: Fear of failure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Investigators plan to use the double-blind procedure, as neither therapists will be informed about the arm (arms will be coded in the scripts), nor participants will be informed about conditions in the study, the research hypotheses will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imagery Rescripting with memory reconsolidation disruption (ImRs-DSR) (Experimental): Before treatment each participant took part in two imagery sessions during which a cognitive-behavioral therapist (CBT) asked him/her to recall three events of being criticized for failures (2 past and 1 future events). The treatment scenario involved memory anticipation (similarly framed for all scenarios) that required recalling three images one after another: the image of self, the surroundings, and the person of the critic involved in the scene.
  After 10 minute break (reconsolidation disruption window) the imagery of the critic was followed by the rescripting part, in which: 1) the therapist enters the scene and prevents the criticism 2) the therapist addresses a critic and points out the child's needs 3) the therapist addresses the child and acknowledges its needs 4) the therapist suggests to the child to perform an activity that would meet its needs.
  Interventions: Behavioral: ImRs-DSR
- Imagery Rescripting regular (ImRs) (Active Comparator): Before treatment each participant took part in two imagery sessions during which a cognitive-behavioral therapist (CBT) asked him/her to recall three events of being criticized for failures (2 past and 1 future events). The treatment scenario involved memory anticipation (similarly framed for all scenarios) that required recalling three images one after another: the image of self, the surroundings, and the person of the critic involved in the scene.
  Immediately after the imagery of the critic the rescripting part was presented, in which: 1) the therapist enters the scene and prevents the criticism 2) the therapist addresses a critic and points out the child's needs 3) the therapist addresses the child and acknowledges its needs 4) the therapist suggests to the child to perform an activity that would meet its needs.
  Interventions: Behavioral: ImRs

INTERVENTIONS:
Behavioral: ImRs-DSR — Imagery Rescripting with Memory Reconsolidation Disruption
  Arms: Imagery Rescripting with memory reconsolidation disruption (ImRs-DSR)
Behavioral: ImRs — Imagery Rescripting regular
  Arms: Imagery Rescripting regular (ImRs)

SUMMARY:
This clinical trial compares the effects of Imagery Rescripting intervention with and without memory reconsolidation disruption procedure (ImRs-DSR and ImRs accordingly), to provide evidence for the superiority of the ImRs-DSR. Tested effects include a decrease in psychophysiological (Skin Conductance Level, Salivary alpha amylase) and subjective (questionnaires & rating) measures in response to imagery scenarios of criticism after 2 weeks of intervention, at 3 & 6-month follow-ups; also, procedures from basic behavior studies (spontaneous recovery, renewal, reinstatement) will be tested; also, generalizability for the imagery of past criticism scenario that wasn't undergoing intervention & novel scenario of future criticism (which would be presented at post-treatment, but not at pre-treatment session) will be tested. The scientific team will recruit a subclinical sample of 48 subjects per group (aiming for the recruitment of 67 subjects due to the high drop-out ratio).

DETAILED DESCRIPTION:
The primary objective of this randomized controlled trial is to compare the Imagery Rescripting intervention with and without memory reconsolidation disruption procedure (ImRs-DSR and ImRs accordingly), to provide evidence for the superiority of the ImRs-DSR on a subclinical sample of at least 96 participants (planned recruitment involves 134 participants to accommodate for drop-outs). Investigators plan to test intervention efficacy by measuring response to imagery scenarios of criticism based on interviews with therapists, conducted before the start of the experiment.

The study uses a 2 x 8 mixed factorial design with two interventions (Imagery Rescripting with and without memory reconsolidation disruption), and 8 time points (pre-treatment (time point 1, TP1), 4 intervention sessions (TP2-TP5), post-treatment after 2 weeks of intervention (TP6), 3- and 6-month follow up (TP7, TP8)). The primary intervention lasts 2 weeks and involves 4 intervention sessions.

In terms of hypotheses, investigators expect that the two-week treatment will result in a stable reduction in subjective and physiological measures of emotional distress related to criticism/failure and ImRs-DSR will be more effective than ImRs in achieving this stability. Herewith, investigators expect that psychophysiological response (sAA and SCL) to the imagery of an autobiographical scenario of being criticized that is used for treatment would drop after treatment when investigated in a familiar context in both groups (H1), and the change will be more pronounced in the superior, i.e. ImRs-DSR group (H2). Investigators hypothesize that after treatment, subjective ratings of negative emotional experience during the treated criticism scenario would also be smaller than before in both groups (H3), however, the decrease will be higher in ImRs-DSR (H4). Investigators also hypothesize that similar effects as those defined in H1 and H3 will be also observed after the presentation of the most aversive part of the scenario (hotspot) i.e. at reinstatement (H5) and that they will be more pronounced in ImRs-DSR (vs ImRs) group (H6). According to our assumptions investigators expect that changes achieved after rescripting one criticism-related scenario in a specific context will generalize to other scenarios (i.e. imagining of untreated past criticism or future criticism scenarios, see Imagery stimuli & interventions section) (H7) and other contexts such as imaging the treated scenario in an unknown room (i.e. renewal) (H8) or various situations verified by PFAI (H9), however, this generalizability will be higher in the ImRs-DSR group with regard to other scenarios (H10), renewal (H11) and PFAI scores (H12). Investigators expect that the changes in reaction (presented in H1, H3, H5, H7, H8, and H9) will be observed after 3 and 6 months (H13), however, a higher decrease will be observed in the ImRs-DSR group (H14).

Primary and secondary outcomes are assessed for criticism-related scenarios using psychophysiology (Skin Conductance Level at pre-, during, and post-treatment, as well as during 3- and 6-month follow-up; Salivary Alpha-Amylase at pre- and post-treatment) and subjective data (online questionnaires and rating, at screening, pre-, during, post-treatment, as well as during 3- and 6-month follow up). Investigators plan to use spontaneous recovery, renewal, and reinstatement procedures to test the efficacy (stability and generalizability) of the studied interventions. For generalizability investigators also plan to test reactions to various imagery scenarios of criticism (un-treated criticism, future criticism). Investigators plan to use 3- and 6-month follow-ups to test long-term effects. Investigators plan to conduct analyses using 2 (arms) x 2 (time points) ANOVA models to check the intervention effects (TP1-TP6 short-term, TP1-TP7/TP8 long-term) on various procedures (spontaneous recovery, renewal, reinstatement). Additional analyses utilize standard NHST calculations and procedures (such as t-tests and correlation coefficients) alongside the conventional ⍺=.05 level.

Investigators plan to use the double-blind procedure, as neither therapists/experimenters will be informed about the arm (arms will be coded in the scripts), nor participants will be informed about conditions in the study, and the research hypotheses will be masked.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-35
* high fear of failure
* not currently undergoing psychotherapy or psychopharmacotherapy
* no severe punitive experiences in the past

Exclusion Criteria:

* current severe affective disorders
* current severe anxiety
* current severe personality disorders
* active suicidality
* psychosis
* substance abuse

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The Performance Failure Appraisal Inventory | Screening, 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  The Performance Failure Appraisal Inventory (PFAI; Conroy, 2001, Polish translation: Golińska, 2017) was used to assess fear of failure. It is a 35-item questionnaire that measures the strength of subjective beliefs about the consequences of failure. The PFAI has five subscales: fear of experiencing shame and embarrassment; fear of devaluing one's self-esteem; fear of having an uncertain future; fear of important others losing interest, and fear of upsetting important others, with scores ranging 35-175.
Subjective ratings at the end of all sessions | Pre-Treatment (TP1), during 2-weeks treatment (TP2-TP5), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Subjective ratings at the end of all sessions- participants were asked to evaluate each fragment of the presented scenarios according to several measures: immersion, focus, emotions (happiness, sadness, guilt, fear, anger, disgust) on a 9-point Likert scale (very low-very high), and valence (very negative-very positive), scores ranging 1-9 for each factor.
SCL recordings | Pre-Treatment (TP1), during 2-weeks treatment (TP2-TP5), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Skin conductance level (SCL) was collected during the audio-guided scenarios' imagery at pre-treatment, treatment, post-treatment, and follow-up sessions. SCL was acquired using Biopack MP160 EDA-MRI system, with a sampling frequency of 2000Hz. The signal was resampled into 1000Hz, then smoothed with median (100 samples), and filtered with a high-passed 1Hz filter. We calculated normalized change in SCL with equation 100✕(SCLStim-SCLbaseline/SCLbaseline), where SCLStim is the mean signal value during the stimulus and SCLbaseline is an SCL reaction during the baseline preceding the first part in each scenario (Sugimine et al., 2020). Our primary outcome was SCL during the imagery of different scenarios, separated for anticipation and hotspot parts.
Saliva sampling sAA | Pre-Treatment (TP1), 2-weeks post-treatment (TP6)
  Saliva samples were collected on pre- and post-treatment with cotton rolls. Samples were collected using cotton rolls that were chewed for 1 min and were later secured in sterile V-bottom tubes and stored at 4°C temperature upon analysis. Samples were coded and sent to the Institute of Human Genetics Polish Academy of Science where the level of alpha amylase was measured.

SECONDARY OUTCOMES:
Beck Depression Inventory | Screening, 6-month Follow-up
  Beck Depression Inventory second edition (BDI-II; Beck, Steer, & Brown, 2005; Polish translation: Łojek & Stańczak, 2019) BDI-II is a self-report scale using 21 items regarding the presence and strength of depression symptoms, with scores ranging 0-63.
Yale-Brown Obsessive-Compulsive | Screening, 6-month Follow-up
  Yale-Brown Obsessive-Compulsive self-report severity scale Y-BOCS-SR (Goodman et al., 1989; Polish translation: translation made by the authors using a standard back-translation method, 2020) a 10-item, self-report questionnaire created to evaluate OCD severity, scores ranging 0-40.
The Alcohol Use Disorders Identification Test | Screening, 6-month Follow-up
  The Alcohol Use Disorders Identification Test AUDIT (Saunders et al., 1993; Polish translation: Babor et al., 1998) is a self-reported tool containing 10 items used to assess recent alcohol consumption, alcohol dependence symptoms, and problems related to alcohol consumption, with scores ranging 0-40.
Drug Abuse Screen Test | Screening, 6-month Follow-up
  Drug Abuse Screen Test DAST 10 (Skinner, 1982; Polish translation: translation made by the authors using a standard back-translation method, 2020) is a self-reported questionnaire to detect drug use disorders, scores ranging 0-10.
DSM Scales | Screening, 6-month Follow-up
  DSM Scales (Craske et al., 2013, own translation); is a set of brief dimensional self-rating questionnaires for social anxiety disorder, agoraphobia, panic disorder, generalized anxiety disorder, and Post Traumatic Stress Symptoms (American Psychiatric Association, 2013, Polish translation: translation made by the authors using a standard back-translation method, 2020). Each scale consists of 10 items relating to the thoughts, feelings, and behaviors the subjects have experienced in the last 7 days. The answers are marked on a 4-point Likert scale (0=never, 4=all the time), with scores ranging 0-4.
Structured Clinical Interview for DSM-5 (SCID-5-PD) | Screening
  Structured Clinical Interview for DSM-5 SCID-5-PD (First et al., 2016, Polish translation: Zawadzki, 2017) is a semistructured clinical interview that evaluates DSM-5 personality disorders under three clusters of A, B, and C, and other specific personality disorders. Based on positive answers to questions clinician diagnose adequate personality disorders.
M.I.N.I. Mini International Neuropsychiatric Interview | Screening
  M.I.N.I. Mini International Neuropsychiatric Interview (Sheehan, et al., 1998, Polish translation: Masiak & Przychoda, 1998) is a short structured interview for DSM IV and ICD 10 disorders, used to assess mental disorders: major depressive disorder, dysthymic disorder, suicidality, mania, panic disorder, agoraphobia, social phobia, specific phobia, obsessive-compulsive disorder, post-traumatic stress disorder, alcohol dependence/abuse, drug dependence/abuse, antisocial personality disorder. Based on positive answers to questions clinician diagnose adequate disorders.
Liebowitz Social Anxiety Scale | Pre-Treatment (TP1), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Liebowitz Social Anxiety Scale (LSAS; Liebowitz, 1987) is a 24-item scale to evaluate fear and avoidance in social situations such as social interaction, public speaking, being observed by others, eating and drinking in public, with scores ranging from 0 to 144.
Pure Procrastination Scale | Pre-Treatment (TP1), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Pure Procrastination Scale (PPS; Steel, 2010; Polish adaptation by Cieciuch and Stępień, with alternations introduced by Stępień and Topolewska, 2014, pp. 152-154) is composed of 12 items, which measures three components of procrastination: decisional delay, implemental delay and delays in lateness/timeliness, with scores ranging 12-60.
Frost Multidimensional Perfectionism Scale | Pre-Treatment (TP1), 2-weeks post-treatment (TP6), 3- & 6-month follow-up (TP7, TP8)
  Frost Multidimensional Perfectionism Scale (Frost MPS; Stöber, 1998; Polish translation: Piotrowski and Bojanowska, 2021) was used to assess overall perfectionism and its dimensions: Personal Standards, Organization, Concern Over Mistakes, Doubts About Actions, Parental Expectations, and Parental Criticism, with scores ranging 35-175.

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław Michałowski, PHD, Principal Investigator — SWPS University
Locations (1):
- SWPS University, Warsaw, Mazowsze, Poland

REFERENCES:
- [Background] Agren T, Engman J, Frick A, Bjorkstrand J, Larsson EM, Furmark T, Fredrikson M. Disruption of reconsolidation erases a fear memory trace in the human amygdala. Science. 2012 Sep 21;337(6101):1550-2. doi: 10.1126/science.1223006. PMID 22997340
- [Background] Arntz A, Weertman A. Treatment of childhood memories: theory and practice. Behav Res Ther. 1999 Aug;37(8):715-40. doi: 10.1016/s0005-7967(98)00173-9. PMID 10452174
- [Background] Conroy, D. E., Willow, J. P., & Metzler, J. N. (2002). Multidimensional fear of failure measurement: The performance failure appraisal inventory. Journal of applied sport psychology, 14(2), 76-90.
- [Background] Morina N, Lancee J, Arntz A. Imagery rescripting as a clinical intervention for aversive memories: A meta-analysis. J Behav Ther Exp Psychiatry. 2017 Jun;55:6-15. doi: 10.1016/j.jbtep.2016.11.003. Epub 2016 Nov 9. PMID 27855298
- [Background] Schiller D, Kanen JW, LeDoux JE, Monfils MH, Phelps EA. Extinction during reconsolidation of threat memory diminishes prefrontal cortex involvement. Proc Natl Acad Sci U S A. 2013 Dec 10;110(50):20040-5. doi: 10.1073/pnas.1320322110. Epub 2013 Nov 25. PMID 24277809
- [Background] Siegesleitner M, Strohm M, Wittekind CE, Ehring T, Kunze AE. Improving imagery rescripting treatments: Comparing an active versus passive approach. J Behav Ther Exp Psychiatry. 2020 Dec;69:101578. doi: 10.1016/j.jbtep.2020.101578. Epub 2020 Jun 9. PMID 32569854
- [Background] Wild J, Clark DM. Imagery Rescripting of Early Traumatic Memories in Social Phobia. Cogn Behav Pract. 2011 Nov;18(4):433-443. doi: 10.1016/j.cbpra.2011.03.002. PMID 22298942
- [Background] Sugimine S, Saito S, Takazawa T. Normalized skin conductance level could differentiate physical pain stimuli from other sympathetic stimuli. Sci Rep. 2020 Jul 2;10(1):10950. doi: 10.1038/s41598-020-67936-0. PMID 32616939
- [Background] First, M. B., Williams, J. B., Karg, R. S., & Spitzer, R. L. (2016). User's guide for the SCID-5-CV Structured Clinical Interview for DSM-5® disorders: Clinical version. American Psychiatric Publishing, Inc..
- [Background] Craske MG, Kircanski K, Epstein A, Wittchen HU, Pine DS, Lewis-Fernandez R, Hinton D; DSM V Anxiety; OC Spectrum; Posttraumatic and Dissociative Disorder Work Group. Panic disorder: a review of DSM-IV panic disorder and proposals for DSM-V. Depress Anxiety. 2010 Feb;27(2):93-112. doi: 10.1002/da.20654. PMID 20099270